CLINICAL TRIAL: NCT01688193
Title: Randomized, Open, 2-way Cross Over, Single Dose Study to Evaluate and Compare Safety and Pharmacokinetics of the HCP1004 and VIMOVO 500/20mg in Healthy Korean Male
Brief Title: Study to Evaluate and Compare Safety and Pharmacokinetics of the HCP1004 and VIMOVO 500/20mg in Healthy Korean Male
Status: Completed | Type: Observational
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: HM-ESNP-102
Record Dates: First submitted 2012-09-14; First posted 2012-09-19 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2013-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HCP 1004
- Vimovo 500/20mg

SUMMARY:
The purpose of this study is to Evaluate and Compare Safety and Pharmacokinetics of the HCP1004 and VIMOVO 500/20mg in Healthy Korean Male

ELIGIBILITY:
Inclusion Criteria:

* BMI: 18.0 - 27.0 kg/m2
* Willingness to sign the written Informed Consent Form

Exclusion Criteria:

* Evidence of clinically relevant pathology
* History of relevant drug and food allergies
* Positive screen on drugs of abuse
* Participation in a drug study within 60 days prior to drug administration.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy korean male
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2012-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
AUClast, Cmax of Naproxen and Esomeprazole | Naproxen : 0h,30min, 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, 72h, Esomeprazole : 0h, 10min, 20min, 30min, 45min, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12h

SECONDARY OUTCOMES:
Tmax, t1/2, CL/F, AUCinf of Naproxen and Esomeprazole | Naproxen : 0h, 30min, 1, 2, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, 72h Esomeprazole: 0h, 10min, 20min, 30min, 45min, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12h

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Wang-Smith L, Fort J, Zhang Y, Sostek M. Pharmacokinetics and relative bioavailability of a fixed-dose combination of enteric-coated naproxen and non-enteric-coated esomeprazole magnesium. J Clin Pharmacol. 2012 May;52(5):670-80. doi: 10.1177/0091270011405500. Epub 2011 May 31. PMID 21628602